CLINICAL TRIAL: NCT02036411
Title: Does Clomiphene Citrate Used for Induction of Ovulation Effect Levels of AMH and Inhibin B
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Taner A Usta, MD, MD, Bagcilar Training and Research Hospital
Other Study IDs: BEH GynObs-5
Record Dates: First submitted 2013-10-10; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: clomiphene citrate; amh; inhibin b
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
100mg clomiphene citrate used for ovulation induction. The investigators take blood sample at 3 and 10 days of menstruation and count AMH and inhibin B.

DETAILED DESCRIPTION:
100mg clomiphene citrate used for ovulation induction. The investigators take blood sample at 3 and 10 days of menstruation. AMH and inhibit B level will be measured in serum. We want to search relation of AMH, inhibin b and ovulation induction.

ELIGIBILITY:
Inclusion Criteria:

* Infertility treatment

Exclusion Criteria:

* Previous ovarian surgery
* Single functioning ovary

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women receiving infertility treatment
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Does Clomiphene Citrate Used for Induction of Ovulation Effect Levels of AMH level | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: TANER USTA, M.D, Principal Investigator — Bagcilar Training and Research Hospital, Istanbul, Turkey.
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)